CLINICAL TRIAL: NCT05517967
Title: An Examination of Brown Adipose Tissue and Energy Expenditure in Infants
Acronym: Born2Burn
Status: Recruiting | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Emily W. Flanagan, MS, PhD, Postdoctoral Researcher, Women's Health, Pennington Biomedical Research Center
Other Study IDs: PBRC 2021-054
Record Dates: First submitted 2022-08-24; First posted 2022-08-26 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Cold Induced Thermogenesis
Keywords: Infant; Energy Expenditure; Indirect Calorimetry; Brown Fat; Neonatal; Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Human milk, if applicable
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Excess fetal adipose tissue growth during intrauterine development increases future obesity risk. Development of brown adipose tissue, a highly thermogenic organ in utero, may affect postnatal energy expenditure, thus influencing obesity risk. This pilot research study is designed to understand the developmental origins of energy balance by examining maternal and neonatal factors that influence neonatal brown adipose tissue and to quantify its physiological relevance to energy expenditure in human neonates.

DETAILED DESCRIPTION:
The developmental origins of obesity begin in utero with growth and differentiation of adipose tissue. Fetal white adipose tissue accretion is highly variable and dependent on the maternal intrauterine environment. Unlike white adipose tissue, brown adipose tissue has a high capacity for thermogenesis. Brown adipose tissue is present at birth and it is believed to support the critical function of thermoregulation in early postnatal life. Therefore, Brown adipose tissue may also influence the development of neonatal energy balance. Similar to white adipose tissue, it is hypothesized that development of Brown adipose tissue in utero is also influenced by maternal factors such as prepregnancy body mass index and gestational weight gain. The research aims of this study to 1) identify maternal and neonatal factors that contribute to neonatal Brown adipose tissue and 2) to identify changes in neonatal Brown adipose tissue and to energy expenditure in response to a mild cold exposure. To achieve these aims, we will conduct a pilot and feasibility study that is cross-sectional, observational study in up to 60 infants 0-3 weeks of age. Using state-of-the-art methodology, we will assess brown adipose tissue, body composition, and resting metabolic rate under thermoneutral and mild-cold stimulated conditions.

ELIGIBILITY:
Inclusion Criteria:

* aged 0 weeks to less than 3 weeks at visit 1
* be willing to complete MRI procedures

Exclusion Criteria:

* Unable to complete two clinic visits within 14 days
* Born with health conditions that would render the procedures unsafe
* Born earlier than 36 and 0 days gestation
* Taken a steroid drug since birth
* Implanted metal or electronic objects that render MRI unsafe

Max Age: 5 Weeks | Sex: All
Age Groups: Child
Study Population: This study will enroll neonates from two mechanisms: 1) recruited from the greater Baton Rouge area, and 2) recruited from an ongoing prenatal weight maintenance intervention randomized controlled trial (R01DK099175).
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-08-17 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Brown Adipose Tissue Fat-signal Fraction Difference Between Thermoneutral and Mild-Cold Environment | 14 days
  The difference in the infants' fat-signal fraction (ratio of lipid to water, expressed as a percentage), assessed by Magnetic Resonance Imaging, between a thermoneutral environment and a mild-cold exposure.
Energy Expenditure Difference Between Thermoneutral and Mild-Cold Environment | 14 days
  The difference in the infants' energy expenditure (expressed as kilocalories per day), assessed by room calorimetry, between a thermoneutral environment and a mild-cold exposure.

CONTACTS AND LOCATIONS:
Overall Officials: Emily W Flanagan, PhD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Flanagan EW, Altazan AD, Carmichael OT, Hu HH, Redman LM. Practical application of in vivo MRI-based brown adipose tissue measurements in infants. Obesity (Silver Spring). 2021 Oct;29(10):1676-1683. doi: 10.1002/oby.23237. PMID 34553508